CLINICAL TRIAL: NCT05099666
Title: A Phase 1b/2 Trial of Lurbinectedin Plus Doxorubicin in Leiomyosarcoma
Brief Title: Lurbinectedin + Doxorubicin In Leiomyosarcoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Gregory Cote, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-437
Record Dates: First submitted 2021-10-01; First posted 2021-10-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Advanced Soft-tissue Sarcoma; Metastatic Soft-tissue Sarcoma; Advanced Leiomyosarcoma; Leiomyosarcoma Metastatic
Keywords: Advanced Soft-tissue Sarcoma; Metastatic Soft-tissue Sarcoma; Advanced Leiomyosarcoma; Leiomyosarcoma Metastatic
MeSH Terms: conditions — Sarcoma | interventions — PM 01183; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lurbinectedin + Doxorubicin Phase I (Experimental): The phase 1b trial will follow a standard 3+3 design. Upon determination of the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of lurbinectedin plus doxorubicin. A treatment cycle will be defined as 21 consecutive days. Treatment will be administered on an outpatient basis
  * Lurbinectedin
  * Doxorubicin
  Interventions: Drug: Lurbinectedin; Drug: Doxorubicin
- Lurbinectedin + Doxorubicin at RP2D (Experimental): The randomized two arm phase 2 trial will begin following the determination of the RP2D for lurbinectedin and doxorubicin.
  * Participants will be randomized 1:1 to enroll to either Arm 1 or Arm 2
  * Participants enrolled to Arm 1 will receive Lurbinectedin with Doxorubicin at the RP2D defined during the phase 1b portion of the trial.
  Interventions: Drug: Lurbinectedin; Drug: Doxorubicin
- Doxorubicin Monotherapy (Active Comparator): The randomized two arm phase 2 trial will begin following the determination of the RP2D for lurbinectedin and doxorubicin.
  * Participants will be randomized 1:1 to enroll to either Arm 1 or Arm 2
  * Participants enrolled to Arm 2 will receive Doxorubicin at the standard dose of 75 mg/m2
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Lurbinectedin — Dosage per protocol, escalation per protocol, IV over 60 minutes (± 5 minute infusion window), schedule per protocol
  Other Names: Zepzelca
  Arms: Lurbinectedin + Doxorubicin Phase I; Lurbinectedin + Doxorubicin at RP2D
Drug: Doxorubicin — Dosage per protocol, IV per institutional standards of practice and the FDA package insert, schedule per protocol
  Other Names: Adriamycin

SUMMARY:
This research study involves the study drug lurbinectedin in combination with doxorubicin.

This research has two parts. The first part is being done to determine the tolerability of lurbinectedin with doxorubicin in people with soft tissue sarcoma. The second part is a randomized study to determine which is more effective at treating leiomyosarcoma, lurbinectedin with doxorubicin or lurbinectedin alone.

DETAILED DESCRIPTION:
This is an open label phase 1b/2 study exploring the safety and efficacy of lurbinectedin with doxorubicin.

- The phase 1b trial will follow a standard 3+3 design. Upon determination of the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of lurbinectedin plus doxorubicin, the randomized phase 2 trial in participants with advanced leiomyosarcoma (LMS) will commence. Participants will be randomized 1:1 for enrollment to one of two treatment arms:

* Arm 1: Lurbinectedin with Doxorubicin
* Arm 2: Doxorubicin Monotherapy

This is a Phase Ib/II clinical trial. A Phase Ib clinical trial tests the safety of an investigational drug combination and also tries to define the appropriate dose of the investigational drugs to use for further studies. "Investigational" means that the drugs are being studied.

The U.S. Food and Drug Administration (FDA) has not approved lurbinectedin for this specific disease but it has been approved for the treatment of small cell lung cancer.

The U.S. FDA has approved doxorubicin as a treatment option for soft-tissue sarcoma.

Lurbinectedin is a synthetically derived chemical that binds to DNA. The binding to DNA likely induces cell death. Doxorubicin is a cytotoxic chemotherapy drug that kills cancer cells by several mechanisms including binding to DNA.

ELIGIBILITY:
Inclusion Criteria:

* For Enrollment to Phase 1b: Participants must have histologically confirmed advanced or metastatic soft-tissue sarcoma and no curative multimodality treatment options available.
* For Enrollment to Phase 2: Participants must have histologically confirmed advanced or metastatic leiomyosarcoma (LMS) and no curative multimodality treatment options available.
* Participants must have measurable disease per RECIST 1.1 criteria
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of lurbinectedin in combination with doxorubicin in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%,).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute Neutrophil Count ≥ 1,500/mcL
  * Hemoglobin (Hgb) ≥ 8 g/dl (transfusion support permitted)
  * Platelet Count ≥ 100,000/mcL
  * Total Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST (SGOT) / ALT(SGPT) ≤ 2.5 × institutional ULN, OR ≤ 5 × institutional ULN if elevation is a result of metastases
  * Creatinine ≤ 1.5 × institutional ULN, OR Creatinine Clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above 1.5 × institutional normal (calculated via the Cockcroft-Gault equation)
  * Creatine Phosphokinase (CPK)< 2.5 × institutional ULN on two different determinations performed one week (± 1 day) apart
* For participants with known chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with known HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Left ventricular ejection fraction (LVEF) ≥ 50% on screening echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
* The effects of lurbinectedin or doxorubicin on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of study agent administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have archival tissue available for analysis in the form of a formalin-fixed paraffin embedded (FFPE) block or unstained slides. Participants without archival tissue available may be enrolled with approval of the Sponsor-Investigator. Note: confirmation of availability of archival tissue is the only requirement for eligibility, archival tissue does not need to be received by the study team or site prior to enrollment.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as assessed by the treating investigator may be included with the approval of the Sponsor-Investigator.

Exclusion Criteria:

* Participants who have received prior anthracycline or trabectedin (Yondelis, ET-743), including prior exposure to doxorubicin or liposomal doxorubicin.
* Participants who have received more than 2 prior lines of cytotoxic chemotherapy for the phase 1b study and no more than 1 prior line of cytotoxic chemotherapy for the phase 2 study. There is no limit on the number of prior lines of non-cytotoxic chemotherapy (e.g., pazopanib, immunotherapy).
* Prior exposure to lurbinectedin (PM01183).
* Participants who have received prior radiation treatment of > 45 Gy to the pelvis.
* Participants who have received or undergone prior chemotherapy within 14 days of cycle 1 day 1, therapeutic radiation therapy within 21 days of cycle 1 day 1 or major surgery within 21 days of cycle 1 day 1.
* Participants who have received prior palliative radiation therapy within 7 days of cycle 1 day 1.
* Participants who have received prior antibody-based therapy (e.g., nivolumab) within 4 weeks or 3 half-lives (whichever is shorter) of cycle 1 day 1.
* Participants who have received prior oral small molecule or tyrosine kinase inhibitor (TKI) therapy within 2 weeks or 3 half-lives (whichever is shorter) of cycle 1 day 1.
* Participants who have not recovered to ≤ Grade 1 or baseline from adverse events attributed to any prior anti-cancer therapy, with the exceptions of alopecia, controlled endocrine toxicity (e.g., hypothyroidism), and cutaneous toxicity which will be permitted at Grade 2.
* Participants who are receiving any other investigational agents.
* Participants with known CNS disease involvement, with the exception of patients with brain metastases that have been previously treated and have remained stable on MRI ≥ 28 days prior to cycle 1 day 1 without use of steroids or anti-epileptic medications.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lurbinectedin or doxorubicin.
* Participants receiving any medications or substances that are strong or moderate inhibitors or inducers of CYP3A, CYP2D6, or P-gp are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the participant must be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic indwelling drains, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of interstitial pneumonitis or pulmonary fibrosis.
* Known cardiomyopathy.
* Pregnant women are excluded from this study because lurbinectedin and doxorubicin are anti-cancer agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lurbinectedin or doxorubicin, breastfeeding must be discontinued if the mother is treated with lurbinectedin or doxorubicin. A negative pregnancy test is required for women of childbearing potential prior to the first dose of study medication.
* Immunocompromised patients, including patients who are known to be seropositive for human immunodeficiency virus (HIV) due to the increased risk of lethal infections when treated with marrow-suppressive therapy. HIV testing is not required as part of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of lurbinectedin with doxorubicin in participants with advanced soft-tissue sarcoma | 21 Days
  The MTD will be defined as the dose where less than 1 in 3 patients experience a DLT. At least 6 patients must be treated at this dose level. DLTs will be defined as toxicities experienced by participants enrolled to the phase 1b portion of the trial that are considered at least possibly related to the treatment regimen, occur during the first cycle of treatment.
PFS rate of lurbinectedin with doxorubicin compared to doxorubicin alone in participants with advanced LMS | Up to 5 years
  Progression-Free Survival (PFS) is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.

SECONDARY OUTCOMES:
Disease Control Rate Phase 1b | 6 Months
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria
Disease Control Rate Phase 1b | 12 Months
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria
Progression Free Survival Phase 1b | Up to 5 years
  PFS is defined as the time from as the time from randomization (or registration) to the earlier of progression or death due to any cause, whichever occurs first
Overall Survival Phase 1b | Up to 5 years
  OS is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Objective Response Phase 1b | Up to 5 years
  assessed by RECIST version 1.1 criteria
Disease Control Rate Phase 2 | 6 Months
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria
Disease Control Rate Phase 2 | 12 Months
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria
Overall Survival Rate Phase 2 | Up to 5 years
  OS is defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Objective Response Rate Phase 2 | Up to 5 years
  assessed by RECIST version 1.1 criteria
Number of Participants Treatment Related Adverse Events | Up to 5 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cote, M.D. Ph.D, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Mayo Arizona, Phoenix, Arizona
  - Mayo Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation